CLINICAL TRIAL: NCT05463406
Title: Procalcitonin and Lung Ultrasonography Based Antibiotherapy in Patients With Lower Respiratory Tract Infection in Swiss Emergency Departments: Pragmatic Stepped-wedge Cluster-randomized Trial
Brief Title: Procalcitonin and Lung Ultrasonography Guided Antibiotherapy in Emergency Departments
Acronym: PLUS-IS-LESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Boillat-Blanco Noemie (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); University Hospital, Basel, Switzerland (Other); Kantonsspital Baden (Other); Hôpital Intercantonal de la Broye, Payerne, Switzerland (Unknown); Réseau Hospitalier Neuchâtelois (Other); Hôpital Riviera-Chablais, Vaud-Valais (Other); Luzerner Kantonsspital (Other); Cantonal Hosptal, Baselland (Other); St. Claraspital AG (Other)
Responsible Party: Sponsor-Investigator, Dr Boillat-Blanco Noemie, Sponsor and National coordinating investigator, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: PLUS-IS-LESS; SNSF 33IC30_201300 (Other Grant/Funding Number: SNSF)
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Lower Respiratory Tract Infection
Keywords: pneumonia; lung ultrasonography; procalcitonin; clinical prediction score; antimicrobial stewardship
MeSH Terms: conditions — Pneumonia | interventions — Algorithms

STUDY DESIGN:
Intervention Model Description: Pragmatic stepped-wedge cluster-randomized controlled clinical trial investigating a new algorithm combining a clinical score, LUS and PCT results (The PLUS algorithm) for the management of LRTIs among adults in EDs. The unit of randomization will be the ED.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The PLUS algorithm (Experimental): The PLUS clinical management algorithm:
  EDs having switched to the intervention period (intervention group) will manage their patients using the PLUS algorithm.
  The PLUS algorithm starts with a validated pneumonia clinical prediction score (score of Van Vugt), followed by LUS. In case of positive results of any of these tests, PCT is measured to identify patients who will most likely benefit from antibiotics. A validated clinical severity score will ensure the safety of the intervention in those with discordant results (LUS consolidation and low PCT).
  Interventions: Other: The PLUS algorithm
- Usual care (Other): Usual care: management as usual
  Interventions: Other: Usual care

INTERVENTIONS:
Other: The PLUS algorithm — Combination of a clinical prediction score and LUS, and if needed PCT measurement
  Arms: The PLUS algorithm
Other: Usual care — Management as usual
  Arms: Usual care

SUMMARY:
Acute respiratory infections are a common reason of attendance at emergency departments. It is also the main reason of unnecessary antibiotic prescription. Antibiotics save lives, but can also directly harm patients by causing antibiotic-associated adverse events. Antibiotic use is directly related to resistance, which is one of the major threats of our century. In addition, some microorganisms live in and on the human body and promote many aspects of our health. Antibiotic treatment can disturb those microorganisms and therefore have long-lasting negative effects on our health.

Unfortunately, it is difficult to differentiate between viral infections, which usually heal spontaneously, and bacterial pneumonia, which needs antibiotics treatment. This is one of the reasons of this over-prescribing of antibiotics.

This project aims to reduce widespread use of antibiotics in the emergency department through a new diagnostic strategy of bacterial pneumonia. This strategy includes sequential use of well-known techniques: a clinical score, lung ultrasound and finally a biomarker, procalcitonin. The latter tends to be higher in bacterial infections. The combination of these different tests improves the diagnostic process and allows improved use of targeted antibiotics, with the ultimate goal of better patient management.

The study will compare the antibiotic prescription rate and the clinical course of patients managed using this new diagnostic approach with those managed as usual. The project will also evaluate the acceptability and feasibility of this strategy and its cost-effectiveness. These two aspects are essential for a wider implementation of this innovative diagnostic approach and decrease antibiotic resistance.

DETAILED DESCRIPTION:
Background Community-acquired lower respiratory tract infections (LRTI) are one of the most common motivations for emergency department (ED) consultations and stands as the leading cause of inappropriate antibiotic prescription. Besides the side effects, antibiotic overuse alters the microbiome and generates antibiotic resistance. When assessing patients with LRTIs, the challenge for ED physicians is to identify those with community-acquired pneumonia (CAP) of bacterial origin, who will most likely benefit from antibiotics. The low diagnostic accuracy of existing tools, as well as the poor adherence of clinicians to test guidance are leading causes of inappropriate antibiotic use.

Several diagnostic tests can assist in identifying patients with LRTI who require antibiotics. Clinical prediction score can refine the probability of CAP. Lung ultrasound (LUS) has a better diagnostic performance than chest X-ray, the historic reference imaging modality to consolidation in ED. LUS is performed quickly at the bedside without radiation. Procalcitonin (PCT) is a host inflammatory biomarker which tends to be higher in bacterial infections. PCT can be used safely to guide antibiotics use, while its impact on prescription is controversial. None of these tools on its own is sufficient to optimize antibiotic prescription, while a combined approach could better guide clinicians.

Rationale The investigators propose to evaluate the use of a decision support tool to guide antibiotics use in the ED as the summative value of LUS with PCT remains unknown in this setting.

Pragmatic stepped-wedge cluster-randomized controlled clinical trial investigating a new algorithm combining a clinical score, LUS and PCT results (The PLUS algorithm) for the management of LRTIs among adults in EDs. The unit of randomization will be the ED.

Primary safety objective To demonstrate non-inferiority of the intervention in terms of clinical failure by day 28.

Co-primary efficacy objective To show a 15% reduction in the proportion of patients with LRTIs prescribed an antibiotic by day 28 in the intervention group compared with the usual care group.

Secondary objectives

1. To compare the quality of life (bothersomeness of CAP-related symptoms) on day 7, day 28 and day 90 between patients in the intervention and control groups.
2. To evaluate the acceptability and feasibility of the intervention through the identification of barriers and facilitators in patients and physicians.
3. To assess the incremental cost-effectiveness of the intervention as compared to usual care using a within-trial (short-term), and a model-based (long-term) economic evaluation.
4. To develop an advanced automatic LUS image analysis method using machine learning to assist in LUS diagnosis and risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients aged 18 years or more
* Acute LRTI (acute illness, less than 21 days, with at least one lower respiratory tract symptom, i.e. cough, sputum, dyspnea, chest pain and no alternative explanation)
* At least one of the following clinical criteria:

  * Focal abnormal auscultation (decreased breath sounds, crackles, bronchial breath sounds)
  * Fever (documented temperature ≥ 38°C in the last 24 hours, including self-measured temperature ≥ 38°C)
  * Tachypnea (respiratory rate ≥ 22/minute)
  * Tachycardia (heart rate ≥ 100/minute)

Exclusion Criteria:

* Previous receipt of a quinolone, macrolide or ceftriaxone or, of more than one dose of any other antibiotic within 72h prior to enrolment (excepted prophylactic antibiotics or antibiotics given for urinary tract infection)
* Previous hospital stay in the last 14 days
* Cystic fibrosis
* Severe COPD (≥GOLD 3 or if not available, as a proxy: exacerbation treated with antibiotics during the last 6 months)
* Severe immunodeficiency (drug-induced neutropenia with <500 neutrophils/mm3, HIV infection with CD4<200 cells/mm3, solid organ or bone marrow transplant recipient, prednisone ≥ 20mg/day for >28 days)
* Initial admission of the patient in the intensive care unit
* Microbiologically-documented SARS-CoV-2
* Incapacity of discernment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | Day 28
  Proportion of patients with clinical failure (defined as a composite of any of the following: death or secondary ICU admission or secondary admission to hospital or hospital re-admission after index hospital discharge or complications due to the LRTI [empyema, lung abscess])
Efficacy outcome | Day 28
  Proportion of patients prescribed an antibiotic in each intervention group between enrolment and day 28

SECONDARY OUTCOMES:
Quality of life measured with the community-acquired pneumonia symptom questionnaire | Day 7, Day 28, Day 90
  Number of points on the community-acquired pneumonia symptom questionnaire as a surrogate marker of quality of life (range 0 to 90; 90 beeing the worse quality of life)
Hospitalisation | Day 0 to Day 90
  Duration of hospitalisation
Efficacy endpoint | Day 90
  Proportion of patients prescribed an antibiotic in each study group between enrolment and day 28 as well as day 90.
Antibiotic side effects and C. difficile infection | Day 0 to Day 28
  Proportion of patients with antibiotic-related side effects and C. difficile infections in each study group.
Emergency department stay | Day 0 to Day 28
  Length of stay in the emergency department in each study group.
Qualitative evaluation | Day 90
  Acceptability and feasibility of the intervention through extensive identification of barriers and facilitators in patients and physicians conducting qualitative semi-structured interviews
Machine learning of Lung ultrasonography (LUS) images and videos | Day 90
  Diagnostic performance for pneumonia (sensitivity, specificity, AUROC) of artificial intelligence LUS interpretation using expert interpretation as gold standard
Economic evaluation | Day 90
  Cost of the intervention as compared to usual care
Clinical gestalt | Day 0
  Diagnostic performance (sensitivity, specificity, AUROC) of the "Clinical gestalt" of the physician in charge of the patient (probability of pneumonia low/intermediate versus high) versus Van Vugt score (1×absence of runny nose+1×breathlessness+1×crackles+1×diminished vesicular breathing+1×raised pulse (>100/min)+1×fever (temperature >37.8°C: probability of pneumonia low/intermediate (score 0-2 ) versus high (score>=3)) to predict LUS-visualized pneumonia

CONTACTS AND LOCATIONS:
Locations (9):
- Switzerland (9):
  - Cantonal hospital of Baden, Baden, Canton of Aargau
  - University Hospital of Basel, Basel, Canton of Basel-City
  - Kantonsspital Baselland, Liestal, Canton of Basel-City
  - Luzerner Kantonsspital, Lucerne, Canton of Lucerne
  - Réseau Hospitalier Neuchâtelois, Neuchâtel, Canton of Neuchâtel
  - Cantonal Hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud
  - Hôpital Intercantonal de la Broye, Payerne, Canton of Vaud
  - Hôpital Riviera-Chablais, Rennaz, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamping DL, Schroter S, Marquis P, Marrel A, Duprat-Lomon I, Sagnier PP. The community-acquired pneumonia symptom questionnaire: a new, patient-based outcome measure to evaluate symptoms in patients with community-acquired pneumonia. Chest. 2002 Sep;122(3):920-9. doi: 10.1378/chest.122.3.920. PMID 12226033
- [Background] Lhopitallier L, Kronenberg A, Meuwly JY, Locatelli I, Mueller Y, Senn N, D'Acremont V, Boillat-Blanco N. Procalcitonin and lung ultrasonography point-of-care testing to determine antibiotic prescription in patients with lower respiratory tract infection in primary care: pragmatic cluster randomised trial. BMJ. 2021 Sep 21;374:n2132. doi: 10.1136/bmj.n2132. PMID 34548312
- [Background] Lhopitallier L, Kronenberg A, Meuwly JY, Locatelli I, Dubois J, Marti J, Mueller Y, Senn N, D'Acremont V, Boillat-Blanco N. Procalcitonin and lung ultrasonography point-of-care testing to decide on antibiotic prescription in patients with lower respiratory tract infection in primary care: protocol of a pragmatic cluster randomized trial. BMC Pulm Med. 2019 Aug 6;19(1):143. doi: 10.1186/s12890-019-0898-3. PMID 31387559
- [Derived] Bessat C, Bingisser R, Schwendinger M, Bulaty T, Fournier Y, Della Santa V, Pfeil M, Schwab D, Leuppi JD, Geigy N, Steuer S, Roos F, Christ M, Sirova A, Espejo T, Riedel H, Atzl A, Napieralski F, Marti J, Cisco G, Foley RA, Schindler M, Hartley MA, Fayet A, Garcia E, Locatelli I, Albrich WC, Hugli O, Boillat-Blanco N; PLUS-IS-LESS study group. PLUS-IS-LESS project: Procalcitonin and Lung UltraSonography-based antibiotherapy in patients with Lower rESpiratory tract infection in Swiss Emergency Departments: study protocol for a pragmatic stepped-wedge cluster-randomized trial. Trials. 2024 Jan 25;25(1):86. doi: 10.1186/s13063-023-07795-y. PMID 38273319